CLINICAL TRIAL: NCT05550909
Title: A Five-arm Trial Comparing Artesunate-amodiaquine and Artemether-lumefantrine-amodiaquine With or Without Single-dose Primaquine to Reduce P. Falciparum Transmission in Mali
Brief Title: Gametocytocidal and Transmission-blocking Efficacy of ASAQ and ALAQ With or Without PQ in Mali
Acronym: NECTAR4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28041
Record Dates: First submitted 2022-09-15; First posted 2022-09-22 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2022-11

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — amodiaquine, artesunate drug combination; Amodiaquine; Primaquine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a single blind randomised controlled trial. The treating physician and staff involved with assessing all laboratory outcomes of the study are blinded, but no placebo will be used. The study pharmacist will be unblinded and responsible for randomisation and treatment administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- artesunate-amodiaquine (ASAQ) (Active Comparator): Subjects will receive artesunate-amodiaquine (ASAQ) daily for 3 days.
  Interventions: Drug: Artesunate-amodiaquine combination
- ASAQ with 0.25mg/kg primaquine (PQ) (Experimental): Subjects will receive artesunate-amodiaquine (ASAQ) daily for 3 days and a single dose of 0.25mg/kg primaquine (PQ) on the first day of ASAQ treatment.
  Interventions: Drug: Artesunate-amodiaquine combination; Drug: Primaquine Phosphate
- Artemether-Lumefantrine (AL) (Active Comparator): Subjects will receive artemether-lumefantrine (AL) twice daily for 3 days.
  Interventions: Drug: Artemether-lumefantrine
- Artemether-Lumefantrine-Amodiaquine (ALAQ) (Experimental): Subjects will receive artemether-lumefantrine (AL) and amodiaquine (AQ) twice daily for 3 days.
  Interventions: Drug: Artemether-lumefantrine; Drug: Amodiaquine
- Artemether-Lumefantrine-Amodiaquine (ALAQ) with 0.25 mg/kg primaquine (PQ) (Experimental): Subjects will receive artemether-lumefantrine (AL) and amodiaquine (AQ) twice daily for 3 days and a single dose of 0.25mg/kg primaquine (PQ) on the first day of ALAQ treatment.
  Interventions: Drug: Primaquine Phosphate; Drug: Artemether-lumefantrine; Drug: Amodiaquine

INTERVENTIONS:
Drug: Artesunate-amodiaquine combination — Tablets containing 50mg/135 mg or 100mg/270 mg of artesunate/amodiaquine will be administered according to weight as per manufacturer guidelines
  Other Names: Camoquin
  Arms: ASAQ with 0.25mg/kg primaquine (PQ); artesunate-amodiaquine (ASAQ)
Drug: Primaquine Phosphate — The single dose of 0.25mg/kg PQ will be administered in an aqueous solution, according to a standard operating procedure (SOP) provided by the manufacturer.
  Other Names: Primaquine
  Arms: ASAQ with 0.25mg/kg primaquine (PQ); Artemether-Lumefantrine-Amodiaquine (ALAQ) with 0.25 mg/kg primaquine (PQ)
Drug: Artemether-lumefantrine — Tablets containing 20 mg artemether and 120 mg lumefantrine will be administered according to weight as per manufacturer guidelines
  Other Names: Coartem
  Arms: Artemether-Lumefantrine (AL); Artemether-Lumefantrine-Amodiaquine (ALAQ); Artemether-Lumefantrine-Amodiaquine (ALAQ) with 0.25 mg/kg primaquine (PQ)
Drug: Amodiaquine — Tablets containing 153 mg of amodiaquine will be administered according to weight, aiming for a dosage of approximately 10 mg (7.7-15.3mg)/kg/day, given once or twice daily (together with artemether-lumefantrine) for three days.
  Arms: Artemether-Lumefantrine-Amodiaquine (ALAQ); Artemether-Lumefantrine-Amodiaquine (ALAQ) with 0.25 mg/kg primaquine (PQ)

SUMMARY:
The purpose of this study is to compare the gametocytocidal and transmission reducing activity of artesunate-amodiaquine (ASAQ) and artemether-lumefantrine-amodiaquine (ALAQ) with and without a single dose of 0.25mg/kg primaquine (PQ). Outcome measures will include infectivity to mosquitoes at 2, 7 and 14 days after treatment, gametocyte density throughout follow-up, and safety measures including haemoglobin density and the frequency of adverse events.

DETAILED DESCRIPTION:
Full protocol available on request

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 10 years and ≤ 50 years
* Absence of symptomatic falciparum malaria, defined by fever on enrolment
* Presence of P. falciparum gametocytes on thick blood film at a density >16 gametocytes/µL (i.e. ≥ gametocytes recorded in the thick film against 500 white blood cells)
* Absence of other non-P. falciparum species on blood film
* Haemoglobin ≥ 10 g/dL
* Individuals weighing < = 80 kg
* No evidence of acute severe or chronic disease
* Written, informed consent

Exclusion Criteria:

* Women who are pregnant or lactating (tested at baseline). Urine and/or serum pregnancy testing (β-hCG) will be used.
* Detection of a non-P. falciparum species by microscopy
* Previous reaction to study drugs / known allergy to study drugs, such as sudden high fevers, shaking or severe sore throat or ulcers in the mouth during treatment with Amodiaquine
* Current eye disease with retinal damage
* Signs of severe malaria, including hyperparasitaemia (defined as asexual parasitaemia > 100,000 parasites / µL)
* Signs of acute or chronic illness, including hepatitis
* The use of other medication (except for paracetamol and/or aspirin), including antacids, other medicines used to treat malaria, abnormal heart rhythm, depression or mental illness or HIV/AIDS, and medicines that have antibiotic/antifungal properties
* Use of antimalarial drugs over the past 7 days (as reported by the participant)
* Clinically significant illness (intercurrent illness e.g., pneumonia, pre-existing condition e.g., renal disease or HIV/AIDS, malignancy or conditions that may affect absorption of study medication e.g., severe diarrhoea or any signs of malnutrition as defined clinically)
* Signs of hepatic injury (such as nausea and/or abdominal pain associated with jaundice) or known severe liver disease (i.e., decompensated cirrhosis, Child Pugh stage B or C)
* Signs, symptoms or known renal impairment
* Clinically significant abnormal laboratory values as determined by history, physical examination, or routine blood chemistries and haematology values (laboratory guideline values for exclusion are haemoglobin < 10 g/dL, platelets < 50,000/μl, White Blood Cell count (WBC) < 2000/μl, serum creatinine >2.0mg/dL, or ALT more than 3 times the upper limit of normal for age.
* Blood transfusion in the last 90 days.
* Known Electrocardiogram (ECG) corrected QT interval of more than 450 ms
* Documented or self-reported history of cardiac conduction problems
* Documented or self-reported history of epileptic seizures

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Change in mosquito infection rate assessed through membrane feeding assays | 2 days (days 0 and 2): 3 day span
  Within person percent change (presented as percent reduction) in mosquito infection rate in infectious individuals from baseline (day 0, pre-treatment) to day 2 post treatment in the ASAQ, ASAQ-PQ, AL, ALAQ and ALAQ-PQ arms.

SECONDARY OUTCOMES:
Change in mosquito infection rate assessed through membrane feeding assays (all timepoints) | 6 days (day 0, day 2, day 7, day 14, day 21, day 28): 28 day span
  Within person percent change (presented as percent reduction) in mosquito infection rate from baseline to all feeding time-points, with comparison within and between arms.
Mosquito infection rate assessed through membrane feeding assays | 6 days (day 0, day 2, day 7, day 14, day 21, day 28): 28 day span
  Mosquito infection rate at all feeding time-points, with comparison within treatment arms compared to baseline, and between arms.
Human infectivity to locally reared mosquitoes assessed through membrane feeding assays | 6 days (day 0, day 2, day 7, day 14, day 21, day 28): 28 day span
  Infectivity to mosquitoes at all feeding time-points, with comparison within treatment arms compared to baseline, and between arms.
Mosquito infection density assessed through membrane feeding assays | 6 days (day 0, day 2, day 7, day 14, day 21, day 28): 28 day span
  Oocyst intensity (in all/all infected mosquitoes) at all feeding time-points, with comparison within treatment arms compared to baseline, and between arms.
Gametocyte infectivity | 6 days (day 0, day 2, day 7, day 14, day 21, day 28): 28 day span
  Infectiousness to mosquitoes for a given gametocyte density (measured as mosquito infection rate/gametocyte) at all feeding time-points, with comparison within treatment arms compared to baseline, and between arms.
Asexual/sexual stage parasite prevalence | 6 days (day 0, day 2, day 7, day 14, day 21, day 28): 28 day span
  Male and female gametocyte prevalence at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms compared to baseline, and between arms.
  Asexual and total parasite prevalence at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms compared to baseline, and between arms.
Asexual/sexual stage parasite density | 6 days (day 0, day 2, day 7, day 14, day 21, day 28): 28 day span
  Male and female gametocyte density at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms compared to baseline, and between arms.
  Asexual and total parasite density at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms compared to baseline, and between arms.
Sexual stage parasite sex ratio | 6 days (day 0, day 2, day 7, day 14, day 21, day 28): 28 day span
  Male and female gametocyte sex ratio (proportion male) at all time-points, determined by microscopy or molecular assays, with comparison within treatment arms compared to baseline, and between arms.
Sexual stage parasite circulation time | 6 days (day 0, day 2, day 7, day 14, day 21, day 28): 28 day span
  Gametocyte circulation time (cumulative), determined by microscopy or molecular assays, compared within and between treatment arms.
Sexual stage parasite area under the curve (AUC) | 6 days (day 0, day 2, day 7, day 14, day 21, day 28): 28 day span
  Gametocyte area under the curve (cumulative), determined by microscopy or molecular assays, compared within and between treatment arms.
Haemoglobin density | 7 days (day 0, day 1, day 2, day 7, day 14, day 21, day 28): 28 day span
  Haemoglobin density (g/dL) at all time-points, with comparison within treatment arms compared to baseline, and between arms.
Change in haemoglobin density | 7 days (day 0, day 1, day 2, day 7, day 14, day 21, day 28): 28 day span
  Within person percent change (presented as percent reduction) in haemoglobin density (g/dL) from baseline to all time-points, with comparison within and between arms.
Incidence of adverse events | 7 days (day 0, day 1, day 2, day 7, day 14, day 21, day 28): 28 day span
  The frequency and prevalence of adverse events (all AE's, treatment related AE's, and haematological AE's) observed up to and including day 2, 7, and 14 post-treatment, and at all timepoints.

OTHER OUTCOMES:
Parasite genomic and transcriptomic variation assessed in RNA | 6 days (day 0, day 2, day 7, day 14, day 21, day 28): 28 day span
  Parasite genotype and transcriptional analysis at baseline and at post-treatment timepoints.
The impact of plasma biomarkers on malaria transmission efficiency | 6 days (day 0, day 2, day 7, day 14, day 21, day 28): 28 day span
  Plasma biomarkers (antibodies and parasite protein) at baseline and at post-treatment timepoints.
Human genomic variation analysis and association with parasite measure | day 0
  Human genotype analysis at baseline (G6PD, CYP2D6, and HBB type)
ALT/AST/Creatine density | 7 days (day 0, day 1, day 2, day 7, day 14, day 21, day 28): 28 day span
  ALT/AST/Creatine density at all time-points with comparison within treatment arms compared to baseline, and between arms.
Impact of magnetic-activated cell sorting (MACS) enrichment of gametocytes on malaria transmission efficiency | 2 days (day 0, day 2): 3 day span
  • Gametocyte density, mosquito infection rate and mean oocyst intensity before and after MACS, for within treatment arm comparison to baseline and comparison between treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Alassane Dicko, Principal Investigator — Malaria Research and Training Centre, Mali
Locations (1):
- Malaria Research and Training Centre, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No
Anonymised individual participant data may be shared on a digital repository or upon reasonable request.

REFERENCES:
- [Derived] Mahamar A, Vanheer LN, Smit MJ, Sanogo K, Sinaba Y, Niambele SM, Diallo M, Dicko OM, Diarra RS, Maguiraga SO, Youssouf A, Sacko A, Keita S, Samake S, Dembele A, Teelen K, Dicko Y, Traore SF, Dondorp A, Drakeley C, Stone W, Dicko A. Artemether-lumefantrine-amodiaquine or artesunate-amodiaquine combined with single low-dose primaquine to reduce Plasmodium falciparum malaria transmission in Ouelessebougou, Mali: a five-arm, phase 2, single-blind, randomised controlled trial. Lancet Microbe. 2025 Feb;6(2):100966. doi: 10.1016/j.lanmic.2024.100966. Epub 2024 Dec 17. PMID 39701119

DOCUMENTS (1):
  • Study Protocol (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT05550909/Prot_000.pdf